CLINICAL TRIAL: NCT05048121
Title: Multicentric, Randomized, Placebo Controlled, Intra-subject, Double Blind Study to Evaluate the Moisturizing Efficacy of a Dermo-cosmetic Product (CLS02021) Versus a Standard Moisturizer During a 4-week Application Period in Healthy Subjects
Brief Title: RCT to Evaluate the Cosmetic Efficacy of Demo-cosmetic Active Ingredient CLS02021
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anbiome Labs LLC (Other)
Collaborators: Sarajevo School of Science and Technology, Medical School Department (Unknown); Public Institution Sarajevo Pharmacies (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RCT-CLS0521
Record Dates: First submitted 2021-08-27; First posted 2021-09-17 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Overall Skin Appearance; Dry Skin; Eczema
Keywords: Skin Hydration; Cosmetic Appearance; Skin Health; Skin Sensitiviry
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Intervention Model Description: Infra-subject comparisons study. As the study is intraindividual, every subject will apply study product on the one side of the face and placebo on the other side of the face at the same time. Subject will not be aware what product is the study product and application is indicated only by the side of the face products are applied.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, double blind, placebo controlled. All products will be packed in the identical packaging and will be labeled in accordance to randomization technique.
  Label will contain: 4 digit, randomization code of the sample and visible sign "LEFT" or "RIGHT".
  Visible sign ''Left'' or ''Right'' will indicate the side of the face the product will be applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLS02021 - Investigational Product arm (Experimental): Cosmetic cream with proprietary cosmetic ingredient CLS02021.
  Interventions: Other: Cosmetic Active Ingredient CLS02021
- PLC01021 - Placebo Control arm (Placebo Comparator): Cosmetic cream, identical to the studied product but without cosmetic ingredient. Color, texture, scent and the packaging are identical as a IP.
  Interventions: Other: Placebo PLC01021

INTERVENTIONS:
Other: Cosmetic Active Ingredient CLS02021 — Topical, face application of the cream base with the CLS02021, two times a day in a period of 30 days
  Arms: CLS02021 - Investigational Product arm
Other: Placebo PLC01021 — Topical, face application of the cream base, two times a day in a period of 30 days
  Arms: PLC01021 - Placebo Control arm

SUMMARY:
This study will explore the potential of probiotic based, novel cosmetic active ingredient to rebuild the collagen based skin barrier with the overall aim to rejuvenate ageing or damaged skin, improve skin integrity, appearance, beauty, and support personal well-being and vitality.

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects aged 18 to 69 years
2. Subjects who have given and signed written informed consent
3. Subjects who are willing to comply with the study requirements

Exclusion Criteria:

1. Subjects with any systemic disorder or face dermatoses including acne that would in any way confound interpretation of the study results (e.g. atopic dermatitis, eczema, or psoriasis)
2. Subjects with a condition or receiving a medication and/or with a history of medical/surgical events which, in the opinion of the Investigator, could compromise the safety of the subject or affect the outcome of the study
3. Subjects with a history of skin cancer
4. Subjects who have started, stopped or changed of hormonal treatment (contraception, thyroid …) in the 3 months prior the study inclusion
5. Subjects who are sensitive to any compound in the base cream
6. Subjects who are sensitive to any active cosmetic compound including Sphingomielinaze, Hylauronic Acid, Lactic Acid or Lipothecoic acid
7. Subjects who have used systemic drugs for more than 3 consecutive days related to antibiotics, anti-inflammatory, corticoids, anti-acneic in the 4 weeks prior to study inclusion
8. Subjects who have used topical drugs for more than 3 consecutive days related to antibiotics, anti-inflammatory, corticoids, anti-acneic in the 4 weeks prior to study inclusion
9. Subjects who have used scrub, anti-seborrheic topical cosmetic products and/or who have applied self-tanning products on face in the 1 week prior the study inclusion
10. Subjects having applied any topical products on face (including make- up) the day of the study inclusion
11. Subjects who have planned a major surgery during the study requiring hospitalization under general anesthesia and the use of systemic or topical drugs (e.g. antibiotics, anti-inflammatory) for more than 1 week
12. Subjects belonging to the staff of the study center
13. Subjects in an exclusion period or participating in another biomedical research study

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-24 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Moisturizing efficacy | 4 weeks
  Change in Instrument measured hydration and elasticity using corneometry (Bioelectrical Impedance Analysis) on the face from baseline to Week 4 (performed by dermatological examiner-blinded)

SECONDARY OUTCOMES:
Wrinkle depth / Skin quality effect | 4 weeks
  Change in Instrument measured Skin wrinkle depth by photometry (shadow method and picture processing) on the face from baseline to Week 4 (performed by dermatological examiner-blinded)
Sebum production / Skin quality effect | 4 weeks
  Change in Instrument measured Skin greasiness by photometry (sebum production/secretion) on the face from baseline to Week 4 (performed by dermatological examiner-blinded)
Pore size / Skin quality effect | 4 weeks
  Change in Instrument measured Skin pore size by photometry (polarized light and picture processing) on the face from baseline to Week 4 (performed by dermatological examiner-blinded)
Melanin production / Skin quality effect | 4 weeks
  Change in Instrument measured Skin melanin production by photometry (light absorption) on the face from baseline to Week 4 (performed by dermatological examiner-blinded)
Sensitivity / Skin quality effect | 4 weeks
  Change in Instrument measured Skin sensitivity by photometry (light reflection) on the face from baseline to Week 4 (performed by dermatological examiner-blinded)
Pore cleanliness / Skin quality effect | 4 weeks
  Change in Instrument measured Pore cleanliness by photometry (polarized light and picture processing) on the face from baseline to Week 4 (performed by dermatological examiner-blinded)
Self-perceived efficacy | 4 weeks
  Self-perceived efficacy on the skin quality using Efficacy questionnaire at Week 4 as compared to baseline
Sensory evaluation | 4 weeks
  Cosmetic acceptability questionnaire at Week 4
Local Tolerance and Safety | 4 weeks
  Safety and Tolerance, Adverse Events Data Collection by the dermatological examiner

CONTACTS AND LOCATIONS:
Locations (2):
- Bosnia and Herzegovina (2):
  - Medical Department, SSST, Sarajevo
  - Public Institution Sarajevo Pharmacies, Sarajevo

IPD SHARING:
Plan to Share IPD: No